CLINICAL TRIAL: NCT01543399
Title: Vascular Effect of Tibolone Versus Placebo Evaluated by Flow-mediated Dilatation of Brachial Artery
Brief Title: Vascular Effect of Tibolone in the Brachial Artery
Acronym: TDILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selmo Geber (Other)
Responsible Party: Sponsor-Investigator, Selmo Geber, Associate Professor, Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T.FR - 245365; ETIC0417 (Other: ethics committee)
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Menopause
Keywords: Tibolone; climacteric; Doppler; hormone replacement therapy
MeSH Terms: interventions — tibolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tibolone use (Experimental): climacteric women will use Tibolone for 30 days
  Interventions: Drug: Tibolone
- Placebo use (Placebo Comparator): climacteric women will use placebo for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tibolone — Experimental group will use 2.5mg of tibolone for 30 days
  Other Names: Livial
  Arms: Tibolone use
Drug: Placebo — patients of the placebo group will use placebo one a day for 30 days
  Arms: Placebo use

SUMMARY:
The interruption of the secretion of sex steroids occurring during menopause, causes a change in vascular pattern at various levels. As a result, several agencies have side effects that interfere with women's health. The use of hormone replacement therapy has contributed to the improvement in these effects. In previous studies the investigators showed the effect of sex steroids in premenopausal women in the conjugated equine estrogens, medroxyprogesterone acetate and tibolone in menopausal women, on the central retinal arteries. The aim of this study is to evaluate the effects of Tibolone in Flow-Mediated Dilatation of the brachial artery.

DETAILED DESCRIPTION:
Menopause is a transitional phase of the biological evolution of women where there is loss of reproductive capacity. The phenomena are the most striking manifestations represented by vasomotor hot flushes and sweating, the consequent fall in estradiol production by the ovaries. The main landmark of the menopause is menopause, which is the last period governed by the ovaries, reflecting the depletion of the same follicle.

The main clinical manifestations of the climacteric are vascular, acting through mechanisms of action not fully understood. Several studies were published showing its effect on vasomotor tone and demonstrating the production of vasoactive substances by vascular cells induced by them.

The main objective of HRT (Hormone Replacement Therapy), is to improve the physical and psychological state of women who have climacteric disorders, leading to improved quality of life. The American College of Physicians, after careful review of available evidence, it is recommended that all postmenopausal women should be considered eligible to receive HRT and that the decision to treat or not should be individualized. Besides the knowledge of the pattern of endocrine patients climate, the investigators must subject it to full physical examination (pelvic) and exams before planning to start HRT. Complementary tests must be clinically oriented, respecting the resources available. There is no need to make routine use of doses of gonadotropins and sex steroids, which are reserved for certain diagnostic situations where there is any doubt, for example, premature ovarian failure syndrome.

He is currently a world consensus that the best available treatment for menopause is hormone replacement therapy because exogenously resets once the hormones produced by the ovaries. HRT fulfills several objectives: reverse neurovegetative symptoms, improves trophism genital atrophy and genital-urinary, acts in the prevention and treatment of osteoporosis, leading to lower incidence of colorectal cancer, promotes a later onset, lower incidence, evolution and improvement in symptoms of Alzheimer's disease has a positive influence on the view.

The development of HRT and the results that prove their individual benefits and epidemiological brought new questions about the most appropriate way to use the various schemes available. The treatment regimens are designed to establish a hormonal profile similar to that of premenopausal using: estrogens, progestogens and androgens in different doses and routes of administration.

Estrogens are the most commonly used conjugated estrogens. The subcutaneous implants (17 beta estradiol) The percutaneous estradiol in the form of gels, transdermal devices (patches) and Tibolone.

Hormones can be used alone or combined, cyclic or continuous, always trying to individualize each situation in order to provide patients with a regimen that suits your needs and desires.

Since its description in 1989, the extent of dilatation of the brachial artery flow-mediated (FMD) has been used to assess endothelial function. It is believed that ischemia induced by inflation of the cuff cause a dilation of the vessel, leading to an increase in brachial artery flow. This effect seems to be mediated by NO production by normal endothelial cells.

In patients whose bioactivity of NO is decreased or absent on endothelial function impairment, this dilatory response does not happen. The dilation of the brachial artery is thus higher in patients with normal endothelial function than in patients who have a pathology that leads to endothelial injury, among them, Hypertension, Coronary heart disease, diabetes mellitus, smoking, hyperlipidemia and Pre-Eclampsia.

Patients will be randomly divided into two groups of 30, using code envelope with the medication, without her or responsible for the study to know the component to be used (double-blind study), with groups divided as follows:

* Group 1 placebo for 30 days;
* Group 2: Tibolone 2.5 mg / day for 30 days Patients will be evaluated before the use of drugs and the end of their use (28-30 days of medication use).

ELIGIBILITY:
Inclusion Criteria:

* Women without menstrual cycles within the last 12 months and FSH > 30IU/L
* Healthy women
* Women that were not using drugs with potential vascular effect within the last 1 year
* Women that never used hormone replacement therapy

Exclusion Criteria:

* Smoking
* Blood Pressure > 160/90 mm Hg.
* Breast and or endometrial cancer
* History of acute myocardial infarction
* Diabetes
* Vaginal bleeding of any origin
* Hepatic disease
* Thrombophlebitis or thromboembolic disorders

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Diameter measurement of the brachial artery using flow-mediated dilation of post menopausal women, before and after use of tibolone. | 30 days
  We will evaluate the vascular effect of Tibolone on the brachial artery. The diameter of the artery will be measured before and one month after use of Tibolone and, in both situations, before and after the use of a cuff in the forearm. Measurement will be in millimeters.

SECONDARY OUTCOMES:
Patients symptoms before and after the use of Tibolone | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Selmo Geber, MD PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- hospital das Clinicas - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] de Souza MA, de Souza BM, Geber S. Vascular resistance of central retinal and ophthalmic arteries in postmenopausal women after use of tibolone. Menopause. 2012 Mar;19(3):328-31. doi: 10.1097/gme.0b013e3182290b26. PMID 22042323